CLINICAL TRIAL: NCT04333992
Title: A Comparison of Propofol-remifentanil Versus Sevoflurane-remifentanil: the Effect on Acute Postoperative Pain After Total Shoulder Arthroplasty
Brief Title: Propofol Versus Sevoflurane on Acute Postoperative Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yeungnam University College of Medicine (Other)
Responsible Party: Principal Investigator, Eun Kyung Choi, Professor, Yeungnam University College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: KNUH 2016-12-009-001
Record Dates: First submitted 2020-04-01; First posted 2020-04-03 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Postoperative Pain
Keywords: propofol; sevoflurane; anesthesia; shoulder arthroplasty
MeSH Terms: conditions — Pain, Postoperative | interventions — Propofol; Remifentanil; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- propofol-remifentanil group (Active Comparator): Anesthetic induction was achieved with an initial target concentration of propofol 4 ㎍/mL and remifentanil 3-4 ng/mL.
  Anesthesia was maintained with a fixed target concentration of propofol 2-4 ㎍/mL and remifentanil 2-3 ng/mL
  Interventions: Drug: propofol and remifentanil
- sevoflurane-remifentanil group (Active Comparator): Anesthetic induction was achieved with thiopental 5 mg/kg and initial target concentration of remifentanil 3-4 ng/mL.
  Anesthesia was maintained with 1.5-2.5% end-tidal concentration sevoflurane in 50% oxygen with air and remifentanil 2-3 ng/mL
  Interventions: Drug: sevoflurane and remifentanil

INTERVENTIONS:
Drug: propofol and remifentanil — intravenous propofol and remifentanil using target-controlled infusion (TCI) devices
  Arms: propofol-remifentanil group
Drug: sevoflurane and remifentanil — inhalator sevoflurane and remifentanil using target-controlled infusion (TCI) devices
  Arms: sevoflurane-remifentanil group

SUMMARY:
This study was performed to compare the acute postoperative pain intensity and opioid consumption after total shoulder arthroplasty between propofol-remifentanil and sevoflurane-remifentanil anesthesia.

DETAILED DESCRIPTION:
After approval of the Institutional Review Board and written informed consent, 48 patients, aged 18-65 years for shoulder arthroplasty were enrolled in this prospective, randomized, double-blinded study.

Patients were assigned to one of two groups : group PR, the propofol-remifentanil group; and group SR, the sevoflurane-remifentanil group.

In the group PR, anesthetic induction was achieved with an initial target concentration of propofol 4 ㎍/mL and remifentanil 3-4 ng/mL using target controlled infusion (TCI) devices and rocuronium 0.8 mg/kg. After intubation, anesthesia was maintained with fixed target concentration of propofol 2-4 ㎍/mL and remifentanil 2-3 ng/mL to keep acceptable hemodynamic response and bispectral index (BIS) values 40-60.

In the group SR, anesthetic induction was achieved with thiopental 5 mg/kg and initial target concentration of remifentanil 3-4 ng/mL using TCI and rocuronium 0.8 mg/kg. Anesthesia was maintained with 1.5-2.5% end-tidal concentration sevoflurane in 50% oxygen with air and remifentanil 2-3 ng/mL was continuously infused adjusting to maintain an acceptable hemodynamics and BIS values 40-60.

The administration of propofol or sevoflurane with remifentanil was stopped at the surgery ended.

Postoperative pain intensity was assessed using a numerical rating scale (NRS: 0; no pain, 10; worst pain) at the 30 min, 2, 6, 12, 24 h. Also, the patient-controlled analgesia (PCA) was infused immediately after post anesthetic care unit arrival. The PCA device was set to deliver 0.38 ㎍/kg/h of fentanyl as a basal infusion rate and 20 ㎍ on demand with a 15 min lockout time. The total PCA volume, number of patients to need rescue analgesics was recorded.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) I or II and aged 18-65 years for total shoulder arthroplasty

Exclusion Criteria:

* Use of routinely using analgesics, history of neurologic or psychologic disease, body mass index more than 35 kg/m2, and intake of any sedatives or analgesics within 24 h before surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-12-12 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
postoperative pain intensity | 24 hours after surgery
  numerical rating scale 0-10 (NRS: 0; no pain, 10; worst pain)
postoperative opioid consumption | 24 hours after surgery
  total patient controlled anesthesia (PCA) volume

CONTACTS AND LOCATIONS:
Locations (1):
- Eun kyung Choi, Daegu, Korea (the Republic Of), South Korea

IPD SHARING:
Plan to Share IPD: Yes